CLINICAL TRIAL: NCT06702436
Title: Impact of Treatment Approaches on Mortality in Cancer Patients With Non-ST Elevation Myocardial Infarction: Invasive vs. Conservative Strategies
Brief Title: Invasive vs. Conservative Management in Cancer Patients With Non-ST Elevation MI (CAN-NSTEMI)"
Acronym: CAN-NSTEMI
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Arif Timuroğlu, MD, Principal Investigator, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: NONST_MI_ONCOLOGY
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Infarction
Keywords: Non-ST Elevated Myocardial Infarction; Malignancy; Mortality
MeSH Terms: conditions — Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Invasive Treatment Group: The Invasive Treatment Group will include cancer patients aged 18 and older diagnosed with non-ST elevation myocardial infarction (NSTEMI) who received an invasive treatment approach. This group will consist of patients who underwent coronary angiography followed by percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG). These patients may have various cancer types, with no restriction on the diagnosis, but must have been treated with invasive procedures for NSTEMI during their hospitalization. The cohort will be assessed for mortality, re-hospitalization rates, and cardiovascular events. The study will also evaluate factors such as cancer stage, metastasis, and comorbidities to understand the outcomes of invasive treatment in this population.
  Interventions: Other: Observational Study
- Conservative Treatment Group: The Conservative Treatment Group will include cancer patients aged 18 and older diagnosed with NSTEMI and managed with medical treatment alone. This group will consist of patients who received pharmacological management (antiplatelet therapy, anticoagulants, beta-blockers, statins) without coronary angiography or revascularization. These patients may have different cancer types, and the study will focus on those treated conservatively during their hospital stay. Mortality, re-hospitalization, and cardiovascular events will be assessed. The analysis will also consider cancer type, disease stage, comorbidities, and pharmacological therapy's impact on long-term outcomes.
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study — This study does not involve any active intervention. It is an observational study comparing the outcomes of invasive and conservative treatment strategies for non-ST elevation myocardial infarction (NSTEMI) in cancer patients. The treatments are based on the clinical decisions made by the attending physicians

SUMMARY:
This retrospective study investigates the impact of invasive versus conservative management strategies in cancer patients presenting with non-ST elevation myocardial infarction (non-ST MI). Patients aged 18 and older, who were treated for non-ST MI in a hospital setting and had a confirmed cancer diagnosis, are included. The primary outcome is hospital mortality, assessed using GRACE scores to evaluate mortality risk. Patients are grouped based on their received interventions-either invasive (including coronary angiography and revascularization) or pharmacological treatment. Risk factors contributing to mortality, such as cancer type, metastasis presence, comorbidities, and laboratory findings, will also be analyzed to better understand the interplay of oncologic and cardiovascular conditions in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients aged 18 years and older.
* Diagnosis: Patients with a confirmed cancer diagnosis.
* Acute Condition: Patients diagnosed with non-ST elevation myocardial infarction (non-ST MI).
* Treatment: Patients who received either invasive treatment (including coronary angiography and revascularization) or conservative (pharmacological) treatment for non-ST MI.
* Consent: Patients who have provided informed consent or are part of a retrospective study where consent is waived.

Exclusion Criteria:

* Age: Patients younger than 18 years.
* Non-cancer diagnoses: Patients without a cancer diagnosis.
* ST-Elevation Myocardial Infarction: Patients with ST elevation myocardial infarction (STEMI) instead of non-ST elevation myocardial infarction (NSTEMI).
* Pre-existing severe comorbidities: Patients with severe or terminal comorbidities (e.g., end-stage liver disease, end-stage renal disease, or severe cognitive impairment) that would confound the outcomes.
* Incomplete medical records: Patients with missing data on relevant clinical variables (e.g., GRACE score, treatment received, or mortality data).
* Pregnancy: Pregnant patients, as their conditions may complicate the interpretation of results.
* Inability to provide informed consent: Patients unable to provide informed consent (if applicable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients aged 18 and older, diagnosed with cancer and hospitalized for non-ST elevation myocardial infarction (NSTEMI). Both males and females with various cancer types will be eligible, and the study will focus on those receiving either invasive or conservative treatment for NSTEMI. Patients with severe comorbidities, such as end-stage diseases or missing critical data, will be excluded. The study aims to assess the impact of invasive versus conservative treatment strategies on mortality, re-hospitalization, and cardiovascular events in this cohort, which is often underrepresented in clinical trials. This population will help understand optimal treatment approaches for cancer patients with NSTEMI.
Sampling Method: Non-Probability Sample
Enrollment: 12500 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
hospital mortality | From the date of hospital admission for NSTEMI until the occurrence of mortality, cardiovascular events, or hospital discharge, assessed up to 30 days.
  Hospital mortality rate in cancer patients with non-ST elevation myocardial infarction, comparing invasive and conservative treatment strategies

SECONDARY OUTCOMES:
Length of hospital stay: | From the date of hospital admission for NSTEMI until the occurrence of mortality, cardiovascular events, or hospital discharge, assessed up to 100 days.
  Comparison of the duration of hospitalization between the invasive treatment group and the conservative treatment group.
Re-hospitalization rate | The time frame for assessing re-hospitalization is from the date of hospital discharge to 100 days post-discharge
  Rate of readmission after initial discharge, comparing the two treatment strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Arif Timuroğlu, Principal Investigator — ankara oncology trainig and research hospital; İmran Ceren, Principal Investigator — ankara oncology trainig and research hospital
Locations (1):
- Ankara Oncology Training and Research Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No